CLINICAL TRIAL: NCT03923478
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Phase 1b Study to Evaluate the Safety, Efficacy and Mircobiological Response of Oral ABI-M201 in Subjects With Mildly-to-Moderately Active UC With Ongoing Mesalamine Treatment
Brief Title: ABI-M201 in Adult Subjects With Mildly-to-Moderately Active Ulcerative Colitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABI-M201-101
Record Dates: First submitted 2019-04-15; First posted 2019-04-22 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Ulcerative Colitis Chronic Mild; Ulcerative Colitis Chronic Moderate
Keywords: Phase 1B; Randomized; Placebo Controlled

STUDY DESIGN:
Intervention Model Description: Double blind, placebo-controlled trial involving two sequential non-overlapping cohorts, with intervening interim analysis
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ABI-M201 (Experimental): Cohort A: 1 capsule one time a day
  Cohort B: 1- 5 capsules one time a day
  Interventions: Drug: ABI-M201
- Placebo (Placebo Comparator): Cohort A: 1 capsule one time a day
  Cohort B: 1-5 capsules one time a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABI-M201 — Active Treatment
  Arms: ABI-M201
Drug: Placebo — Control Treatment
  Arms: Placebo

SUMMARY:
Phase 1B randomized, double-blind, placebo-controlled, two-cohort clinical trial of ABI-M201 in adult subjects with mildly-to-moderately active Ulcerative Colitis(UC) and ongoing treatment with mesalamine.

DETAILED DESCRIPTION:
This multi-center randomized, double-blind, placebo-controlled study will evaluate the safety of ABI-M201 and its effects on disease activity measures in men and women with mildly-to-moderately active UC and ongoing treatment with mesalamine. The study will consist of 2 sequential, non-overlapping participant cohorts, separated by intervening interim analysis (IA). Both cohorts will involve 8-weeks of study drug treatment. Interim data from the initial treatment cohort (Cohort A) will inform decision to advance to the subsequent second cohort (Cohort B) and its dose selection. 20 subjects will be randomized to cohort A (1:1 allocation) and receive treatment with 1 capsule per day of ABI-M201 versus Placebo. 24 subjects will be randomized to cohort B (3:1 allocation) and receive treatment with up to 5 capsules one time a day of ABI-M201 versus Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of UC for at least 3 months prior to screening, with minimum disease extent of 15 cm from the anal verge
* Mildly to moderately active UC
* Inadequate response to ongoing treatment with oral mesalamine ≥2.4 g/day for ≥4 weeks from screening visit

Exclusion Criteria:

* Possible or confirmed diagnosis of Crohn's Disease or other forms of inflammatory bowel disorders
* Ongoing or failed prior treatment for UC with methotrexate, azathioprine, 6-mercaptopurine, cyclosporine, tofacitinib, mycophenolate mofetil, sirolimus (rapamycin), thalidomide, tacrolimus (FK-506), or biologics (e.g., TNF-alpha-antagonists, anti-integrin therapies, or agents targeting IL-12 or IL-23, etc.)
* Any immunosuppressive condition or treatment with immunosuppressive medications
* History of prior surgical intervention in any region of the gastrointestinal tract (excluding minor surgery)
* Prior diagnosis of any cardiovascular, renal, hepatic, endocrine, infectious, hematological, oncologic, neuro-psychiatric or immune-mediated disorder, which in the opinion of the Principal Investigator might impact the subject's safety or compliance, or the interpretation of results
* Treatment with any other investigational drugs ≤12 weeks prior to baseline visit
* The participant has a condition or is in a situation which, in the Principal Investigator's opinion, may put the participant at significant risk, may confound the study results, or may interfere significantly with the participant's participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 8-weeks
  [Safety]
Incidence of Treatment-Emergent Laboratory Abnormalities | 8-weeks
  [Safety]

SECONDARY OUTCOMES:
Clinical Remission | 8-weeks
  [UC Disease Activity]
Endoscopic Improvement | 8-weeks
  [UC Disease Activity]

CONTACTS AND LOCATIONS:
Locations (11):
- United States (10):
  - (Investigator site), Oakland, California
  - (Investigator Site), San Carlos, California
  - (Investigator Site), Decatur, Georgia
  - (Investigator Site), Shreveport, Louisiana
  - (Investigator Site), Chesterfield, Michigan
  - (Investigator Site), Ypsilanti, Michigan
  - (Investigator Site), Rochester, Minnesota
  - (Investigator Site), Jackson, Tennessee
  - (Investigator Site), Bellevue, Washington
  - (Investigator Site), Milwaukee, Wisconsin
- (Investigator site), Greater Sudbury, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No